CLINICAL TRIAL: NCT00777803
Title: A Prospective, Multicenter, Randomized, Rater- and Subject-Blind, Parallel Group Trial to Investigate the Non-Inferiority of NT 201, Free of Complexing Proteins, in Comparison With Clostridium Botulinum Toxin Type A in the Treatment of Glabellar Frown Lines
Brief Title: NT 201 (Xeomin®/Bocouture®) in Comparison With Clostridium Botulinum Toxin Type A in the Treatment of Glabellar Frown Lines
Acronym: Head2Head
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201 GL_3002; 2008-002713-40 (EudraCT Number)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2012-02-10 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IncobotulinumtoxinA (Xeomin®/Bocouture®) (Experimental): IncobotulinumtoxinA (Xeomin®/Bocouture®), 24 units; mode of administration: intramuscular injection.
  Interventions: Drug: NT 201 (IncobotulinumtoxinA (Xeomin®/Bocouture®))
- OnabotulinumtoxinA (Vistabel®) (Active Comparator): OnabotulinumtoxinA (Vistabel®), 24 units; mode of administration: intramuscular injection.
  Interventions: Drug: OnabotulinumtoxinA (Vistabel®)

INTERVENTIONS:
Drug: NT 201 (IncobotulinumtoxinA (Xeomin®/Bocouture®)) — NT201, also known as IncobotulinumtoxinA (Xeomin®/Bocouture®), active ingredient: Clostridium botulinum neurotoxin type A free from complexing proteins, powder for solution for injection dose, 24 units; one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl). Of the 0.6 mL total injection volume, an aliquot of 0.15 mL was administered in the procerus muscle, aliquots of 0.125 mL were administered in the medial part of the both corrugator muscles and aliquots of 0.1 mL were administered in the middle part of both corrugator muscles.
  Other Names: "Botulinum toxin type A (150 kiloDalton), free from complexing proteins"
  Arms: IncobotulinumtoxinA (Xeomin®/Bocouture®)
Drug: OnabotulinumtoxinA (Vistabel®) — OnabotulinumtoxinA (Vistabel®), active ingredient: Clostridium botulinum neurotoxin type A, powder for solution for injection dose, 24 units; one injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl). Of the 0.6 mL total injection volume, an aliquot of 0.15 mL was administered in the procerus muscle, aliquots of 0.125 mL were administered in the medial part of the both corrugator muscles and aliquots of 0.1 mL were administered in the middle part of both corrugator muscles.
  Other Names: "BOTOX® Cosmetic"; "Botulinum toxin type A (900 kiloDalton)"
  Arms: OnabotulinumtoxinA (Vistabel®)

SUMMARY:
NT 201, also known as IncobotulinumtoxinA (Xeomin®/Bocouture®), is a Botulinum toxin type A preparation free of complexing proteins (150 kiloDalton). Injected into the muscle, NT201 causes a reversible local relaxation of the injected muscle. Botulinum toxin type A is used for aesthetic treatment of mimic wrinkles and in the therapy of neurologic diseases. This study will investigate the safety and efficacy (non-inferiority) of NT 201 in comparison with OnabotulinumtoxinA (Vistabel®) in the treatment of glabellar frown lines.

ELIGIBILITY:
Main Inclusion Criteria:

• Moderate to severe glabellar frown lines at maximum frown (severity score of 2 or 3 on a 4-point facial wrinkle scale) as assessed by the investigator's rating: 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe'.

Main Exclusion Criteria:

* Marked facial asymmetry.
* Ptosis of eyelid and/or eyebrow.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 381 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (17):
- Austria (4):
  - Baden
  - Krems
  - Salzburg
  - Vienna
- Germany (9):
  - Bad Soden
  - Böblingen
  - Cologne
  - Darmstadt
  - Frankfurt
  - Korschenbroich
  - Ludwigshafen
  - Munich
  - Wuppertal
- United Kingdom (4):
  - Glasgow
  - Manchester
  - Suttion Coldfield
  - Winchester

REFERENCES:
- [Result] Sattler G, Callander MJ, Grablowitz D, Walker T, Bee EK, Rzany B, Flynn TC, Carruthers A. Noninferiority of incobotulinumtoxinA, free from complexing proteins, compared with another botulinum toxin type A in the treatment of glabellar frown lines. Dermatol Surg. 2010 Dec;36 Suppl 4:2146-54. doi: 10.1111/j.1524-4725.2010.01706.x. PMID 21134045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized according to a ratio of 3:1 to be either treated with IncobotulinumtoxinA (Bocouture®) or with OnabotulinumtoxinA (Vistabel®).
Period: Overall Study
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Started | 284 | 97
Completed | 269 | 90
Not Completed | 15 | 7
Not completed — Lost to Follow-up | 12 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®) | Total
Number analyzed (Participants) | 284 | 97 | 381
Age Continuous [Mean (Standard Deviation); unit: years] | 41.6 (5.7) | 42.0 (6.0) | 41.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 97 | 381
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder by Independent Rater's Assessment at Maximum Frown at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A subject is a responder if at least 2 out of 3 independent rater identified a response. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 4 weeks thereafter at maximum frown. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 4 weeks after injection
Population: Analysis per protocol: All subjects who received study medication, for whom a facial wrinkle score at maximum frown was observed at baseline and who had no major protocol deviations. Missing facial wrinkle scores were not imputed.
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 93
participants | 267 | 89
Statistical Analysis 1: Comparison: IncobotulinumtoxinA (Xeomin®/Bocouture®) vs OnabotulinumtoxinA (Vistabel®); Null Hypothesis: Response rate of IncobotulinumtoxinA (Xeomin®/Bocouture®) minus the response rate of OnabotulinumtoxinA (Vistabel®) is lower or equal -15% (non-inferiority margin); Test type: Non-Inferiority or Equivalence — A two-sided 95% Newcombe confidence interval for proportions (paired data) was applied. The lower bound of the Newcombe-Wilson confidence interval of the difference in response rates between groups was compared to the non-inferiority margin of -15%; difference of response rates = 0.7, 95% CI 2-sided [-3.2 to 7.1] — Difference of response rates = response rate in IncobotulinumtoxinA (Xeomin®/Bocouture®) - response rate in OnabotulinumtoxinA (Vistabel®)

2. Secondary Outcome: Responder by Independent Rater's Assessment at Maximum Frown at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A subject is a responder if at least 2 out of 3 independent rater identified a response. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 12 weeks thereafter at maximum frown. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 12 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 222 | 73

3. Secondary Outcome: Responder by Independent Rater's Assessment at Rest at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A subject is a responder if at least 2 out of 3 independent rater identified a response. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 4 weeks thereafter at rest. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 4 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 92
participants | 115 | 37

4. Secondary Outcome: Responder by Independent Rater's Assessment at Rest at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A subject is a responder if at least 2 out of 3 independent rater identified a response. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 12 weeks thereafter at rest. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 12 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 100 | 33

5. Secondary Outcome: Responder by Investigator's Assessment at Maximum Frown at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 4 weeks thereafter at maximum frown rated by the investigator. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 4 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 93
participants | 274 | 89

6. Secondary Outcome: Responder by Investigator's Assessment at Maximum Frown at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 12 weeks thereafter at maximum frown rated by the investigator. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 12 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 220 | 76

7. Secondary Outcome: Responder by Investigator's Assessment at Rest at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 4 weeks thereafter at rest rated by the investigator. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 4 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 93
participants | 210 | 66

8. Secondary Outcome: Responder by Investigator's Assessment at Rest at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 12 weeks thereafter at rest rated by the investigator. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 12 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 166 | 51

9. Secondary Outcome: Responder by Patient's Assessment at Maximum Frown at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 4 weeks thereafter at maximum frown rated by the patient. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 4 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 93
participants | 260 | 87

10. Secondary Outcome: Responder by Patient's Assessment at Maximum Frown at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 12 weeks thereafter at maximum frown rated by the patient. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 12 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 202 | 71

11. Secondary Outcome: Responder by Patient's Assessment at Rest at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 4 weeks thereafter at rest rated by the patient. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 4 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 93
participants | 193 | 70

12. Secondary Outcome: Response by Patient's Assessment at Rest at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as an improvement of at least one point on a 4-point facial wrinkle scale from baseline to 12 weeks thereafter rated by the patient. The scale comprises the items 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe' wrinkles.
Time Frame: 12 weeks after injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 152 | 53

13. Secondary Outcome: Responder by Patient's Global Assessment at Week 4
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as a score of at least +2 (moderate improvement) on a 9-point scale (range from +4 complete improvement to -4 very marked worsening) 4 weeks after treatment rated by the patient.
Time Frame: 4 weeks after injection
Population: Analysis per protocol: All subjects who received study medication, for whom a facial wrinkle score at maximum frown was observed at baseline and who had no major protocol deviations. Missing scores were not imputed.
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 277 | 93
participants | 259 | 86

14. Secondary Outcome: Responder by Patient's Global Assessment at Week 12
Description: The Outcome Measure Data Table describes the number of responders. A response is defined as a score of at least +2 (moderate improvement) on a 9-point scale (range from +4 complete improvement to -4 very marked worsening) 12 weeks after treatment rated by the patient.
Time Frame: 12 weeks after injection
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Number analyzed (Participants) | 268 | 88
participants | 229 | 75

ADVERSE EVENTS:
Time Frame: All SAEs/AEs up to 12 weeks after injection.
Description: The table of "Other Adverse Events" includes all non-serious AEs. The investigator asked the patient for AEs systematically at each visit.
Arm/Group | IncobotulinumtoxinA (Xeomin®/Bocouture®) | OnabotulinumtoxinA (Vistabel®)
Serious Adverse Events (participants affected / at risk) | 1/284 | 1/97
Other Adverse Events (participants affected / at risk) | 22/284 | 12/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IncobotulinumtoxinA (Xeomin®/Bocouture®) (N=284) | OnabotulinumtoxinA (Vistabel®) (N=97)
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IncobotulinumtoxinA (Xeomin®/Bocouture®) (N=284) | OnabotulinumtoxinA (Vistabel®) (N=97)
Headache (Nervous system disorders) | 12 | 7
Nasopharyngitis (Infections and infestations) | 11 | 4
Gastrointestinal infection (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 wks before submission. Sponsor to give written opinion within 30 d. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.